CLINICAL TRIAL: NCT01055730
Title: The Impact of Pulmonary Rehabilitation in Interstitial Lung Disease: A Prospective Cohort Study
Brief Title: The Impact of Pulmonary Rehabilitation in Interstitial Lung Disease
Acronym: PR-ILD
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: PR-ILD
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Interstitial Lung Disease
Keywords: Pulmonary rehabilitation; Exercise therapy; Interstitial lung disease; Pulmonary fibrosis; Mobility limitation; Dyspnea; Mental health
MeSH Terms: conditions — Lung Diseases, Interstitial; Pulmonary Fibrosis; Mobility Limitation; Dyspnea; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pulmonary rehabilitation
  Interventions: Other: Pulmonary rehabilitation

INTERVENTIONS:
Other: Pulmonary rehabilitation — Structured education and supervised exercise program, lasting between 6 and 9 weeks.

SUMMARY:
The purpose of this study is to determine if pulmonary rehabilitation has any effect on breathlessness, quality of life, physical function and depression in persons with interstitial lung disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 18 years old) with a diagnosis of ILD who are referred to a participating PR program

Exclusion Criteria:

* Inability to provide informed consent
* Inability to read and write English
* Any other medical condition that significantly limits the subject's ability to perform the functional measures
* Emphysema / Chronic bronchitis (FEV1 / FVC ratio < 60%)
* Previous pulmonary rehabilitation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient with interstitial lung disease who is referred to a participating pulmonary rehabilitation program. These patients typically have exercise limitation and dyspnea, but still possess the ability to perform some exercise.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2010-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
6-minute walk distance | Immediately following completion of pulmonary rehabilitation and 6 months following the start of pulmonary rehabilitation
Quality of life | Immediately following completion of pulmonary rehabilitation and 6 months following the start of pulmonary rehabilitation

SECONDARY OUTCOMES:
Dyspnea | Immediately following completion of pulmonary rehabilitation and 6 months following the start of pulmonary rehabilitation
Depression | Immediately following completion of pulmonary rehabilitation and 6 months following the start of pulmonary rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Harold R Collard, MD, Principal Investigator — University of California, San Francisco; Christopher J Ryerson, MD, Principal Investigator — University of California, San Francisco; Chris Garvey, FNP, Principal Investigator — Seton Pulmonary & Cardiac Rehabilitation
Locations (6):
- United States (5):
  - John Muir Health, Concord, California
  - Seton Pulmonary & Cardiac Rehabilitation, Daly City, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Duke University Medical Center, Durham, North Carolina
  - Inova Fairfax Hospital, Falls Church, Virginia
- University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Ryerson CJ, Cayou C, Topp F, Hilling L, Camp PG, Wilcox PG, Khalil N, Collard HR, Garvey C. Pulmonary rehabilitation improves long-term outcomes in interstitial lung disease: a prospective cohort study. Respir Med. 2014 Jan;108(1):203-10. doi: 10.1016/j.rmed.2013.11.016. Epub 2013 Dec 4. PMID 24332409